CLINICAL TRIAL: NCT00145691
Title: The Effect of Oxcarbazepine in the Treatment of Agitation / Aggression in Dementia (OBAD) - An Eight Week Prospective, Randomized, Double-Blind, Placebo-Controlled, Multi Center Trial. A Phase III Study
Brief Title: The Effect of Oxcarbazepine in the Treatment of Agitation / Aggression in Dementia (OBAD)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Sykehuset Innlandet HF (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: EudraCT number: 2004-005266-20; Sponsor's Protocol Code: 1500
Record Dates: First submitted 2005-09-01; First posted 2005-09-05 (Estimated); Last update posted 2007-03-21 (Estimated); Status verified 2007-03

CONDITIONS: Agitation Aggression in Dementia
MeSH Terms: interventions — Oxcarbazepine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Drug: Oxcarbazepine

SUMMARY:
We intend to conduct a phase III b trial to verify Oxcarbazepine's effect in agitation and aggression in patients with dementia. We designed the study as a randomized, double-blind, placebo-controlled multi center trial. Hundred patients will be included. The treatment period will be eight weeks, with a further follow up of four weeks.

The primary outcome measure will be the reduction in aggression and agitation as measured by means of NPI-NH-subscale agitation / aggression (Neuropsychiatric Inventory, Nursing Home Version). Secondary outcomes are reduction in aggression as measured by BARS (Behavior Agitation Rating Scale)and reduction in the burden to health-care personnel as measured by NPI-NH.

DETAILED DESCRIPTION:
Inclusion criteria: Patients of either gender, 55 years of age or older, living in a nursing home diagnosed with or a strong suspicion of dementia of Alzheimer's type or vascular origin, and BPSD in form of agitation / aggression as measured by subscale of NPI-NH and BARS.

Exclusion criteria: Patients that have any other kind of dementia as FTD, PD or LBD; patients with hepatic or renal failure, or diseases that make it impossible to follow the study schedule; patients on antiepileptics or antipsychotics.

ELIGIBILITY:
Inclusion Criteria:

* Alzheimer's dementia, vascular dementia or mixed forms of both according to ICD10 (F00, F01) criteria.
* The patient is 55 years of age or older.
* Residents at a nursing home and who have been there for at least 4 weeks prior to inclusion.
* Signed informed consent by the patient or the relatives signed agreement that they have no reservations against patient's participation in the study.
* At least one week history of agitation or aggression, score 6 or more in NPI-NH-subscale agitation/aggression.

Exclusion Criteria:

* Previous intolerability or known hypersensitivity to Oxcarbazepine or its equivalents
* Low sodium serum levels <135 mmol/L
* Severe impaired renal function (creatinine clearance <30 ml/min, calculated with Cockroft + Gault's formula)
* Hepatic failure (transaminases (g-GT and ALAT > 3 times upper normal limit).
* Patients with AV-block II and III and all kinds of arrhythmia necessitating a treatment.
* Severe somatic diseases that afford a change of medication and will compromise the attendance to the study.
* Patients on cyclosporine.
* Patients in need of strong analgesics like opioids as codeines
* Patients taking carisoprodol
* Alcohol or drug abuse during the last 12 months (used a higher dosage than prescribed)
* The patient has been on ChEIs or memantine for less than 3 months or any change in the dosage during the last 2 weeks.
* The patient is taking antiepileptics or antipsychotics (may be included two weeks after the use of antipsychotics has been ended).
* The patient is taking MAOI or lithium
* The patient with a dementia of type PDD, FTD or DLB
* The patients with a severe or acute neurological disease (e.g. epilepsy, acute CVE, severe Parkinson's disease, acute confusion) or a severe psychiatric disorder like bipolar disorder, schizophrenia...
* The patients who have participated in another clinical trial during the last 3 months.
* The patients who have been randomized to the same study before.

Min Age: 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100
Dates: Start 2005-09; Study Completion 2006-10 (Actual)

PRIMARY OUTCOMES:
Reduction in aggression and agitation as measured by means of NPI-NH-subscale agitation / aggression (Neuropsychiatric Inventory, Nursing Home Version)

SECONDARY OUTCOMES:
Reduction in aggression as measured by BARS (Behavior Agitation Rating Scale),
Reduction in the burden to health-care personnel as measured by NPI-NH.
Evaluate the concomitant use of acute medication (haloperidol), and compare the frequency and dosage used in the two groups.

CONTACTS AND LOCATIONS:
Overall Officials: Oskar H Sommer, MD, Principal Investigator — Sykehuset Innlandet HF
Locations (1):
- Sykehuset Innlandet HF, Reinsvoll, Oppland, Norway

REFERENCES:
- [Derived] Sommer OH, Aga O, Cvancarova M, Olsen IC, Selbaek G, Engedal K. Effect of oxcarbazepine in the treatment of agitation and aggression in severe dementia. Dement Geriatr Cogn Disord. 2009;27(2):155-63. doi: 10.1159/000199236. Epub 2009 Feb 2. PMID 19182483